CLINICAL TRIAL: NCT06780293
Title: Exploring the Long-term Therapeutic Effects of Laser Acupuncture on Dry Eye and Sjögren's Syndrome-related Dry Eye Symptoms
Brief Title: Laser Acupuncture on Dry Eye and Sjögren's Syndrome-related Dry Eye Symptoms (LADESJS)
Acronym: LADESJS
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Ching-Mao Chang, Director of Division of Integrative Medicine, Center for Traditional Medicine, Taipei Veterans General Hospital, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2024-11-008C
Record Dates: First submitted 2025-01-13; First posted 2025-01-17 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye Syndrome (DES); Laser Acupuncture; Sjögren's Syndrome (SS)
Keywords: Dry eye syndrome; Sjögren's syndrome; Laser Acupuncture; Fengchi (GB20); Zanzhu (BL2); Hegu (LI4); Quchi (LI11)
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: A total of 140 dry eye patients will be recruited and divided into two groups: 70 participants with SJS-DES and 70 with Non-SJS-DES. Participants will be randomly assigned into three groups: Sham+LA group (60 participants receiving 4 weeks of placebo laser acupuncture followed by 4 weeks of active laser acupuncture), LA+LA group (60 participants receiving 4 weeks of active laser acupuncture followed by another 4 weeks of active laser acupuncture), and a Waiting List group (20 participants receiving no laser acupuncture treatment).
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization process will be conducted by a statistical expert using permuted block randomization to generate a "Clinical Trial Randomized Allocation Table." The allocation details will be sealed in envelopes to ensure blinding. Additionally, individual decoding envelopes will be prepared for each participant to allow emergency unblinding without compromising the trial's integrity. The randomization table and grouping details will be securely stored by the statistical expert and the principal investigator, while the individual decoding envelopes will be kept exclusively by the principal investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- LA+LA group of SJS-DES (Experimental): LA+LA group of SJS-DES will receive laser acupuncture at acupoint GB20, BL2, LI4 and LI11 twice a week 8 weeks for efficacy evaluation. And we could use the Numerical Rating Scale (NRS), Schirmer's test, Ocular Surface Disease Index (OSDI), EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI), Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, TCM constitution questionnaire, TCM heart rate variability analysis, nailfold microcirculation assessment, and iris examination for this purpose.
  Interventions: Other: Laser acupuncture (LA); Diagnostic Test: Numerical Rating Scale (NRS); Diagnostic Test: Schirmer's test; Diagnostic Test: Ocular Surface Disease Index (OSDI); Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI); Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) pulse diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) constitution questionnaire; Diagnostic Test: Traditional Chinese Medicine (TCM) heart rate variability analysis; Diagnostic Test: nailfold microcirculation assessment; Diagnostic Test: iris examination
- Sham+LA group of SJS-DES (Sham Comparator): Sham+LA group of SJS-DES will receive sham acupuncture twice a week 4 weeks and then laser acupuncture at acupoint GB20, BL2, LI4 and LI11 twice a week 4 weeks for efficacy evaluation. And we could use the Numerical Rating Scale (NRS), Schirmer's test, Ocular Surface Disease Index (OSDI), EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI), Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, TCM constitution questionnaire, TCM heart rate variability analysis, nailfold microcirculation assessment, and iris examination for this purpose.
  Interventions: Other: Laser acupuncture (LA); Diagnostic Test: Numerical Rating Scale (NRS); Diagnostic Test: Schirmer's test; Diagnostic Test: Ocular Surface Disease Index (OSDI); Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI); Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) pulse diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) constitution questionnaire; Diagnostic Test: Traditional Chinese Medicine (TCM) heart rate variability analysis; Diagnostic Test: nailfold microcirculation assessment; Diagnostic Test: iris examination; Other: Sham Laser Acupuncture
- LA+LA group of Non-SJS-DES (Experimental): LA+LA group of Non-SJS-DES will receive laser acupuncture at acupoint GB20, BL2, LI4 and LI11 twice a week 8 weeks for efficacy evaluation. And we could use the Numerical Rating Scale (NRS), Schirmer's test, Ocular Surface Disease Index (OSDI), EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI), Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, TCM constitution questionnaire, TCM heart rate variability analysis, nailfold microcirculation assessment, and iris examination for this purpose.
  Interventions: Other: Laser acupuncture (LA); Diagnostic Test: Numerical Rating Scale (NRS); Diagnostic Test: Schirmer's test; Diagnostic Test: Ocular Surface Disease Index (OSDI); Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI); Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) pulse diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) constitution questionnaire; Diagnostic Test: Traditional Chinese Medicine (TCM) heart rate variability analysis; Diagnostic Test: nailfold microcirculation assessment; Diagnostic Test: iris examination
- Sham+LA group of Non-SJS-DES (Sham Comparator): Sham+LA group of Non-SJS-DES will receive sham acupuncture twice a week 4 weeks and then laser acupuncture at acupoint GB20, BL2, LI4 and LI11 twice a week 4 weeks for efficacy evaluation. And we could use the Numerical Rating Scale (NRS), Schirmer's test, Ocular Surface Disease Index (OSDI), EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI), Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, TCM constitution questionnaire, TCM heart rate variability analysis, nailfold microcirculation assessment, and iris examination for this purpose.
  Interventions: Other: Laser acupuncture (LA); Diagnostic Test: Numerical Rating Scale (NRS); Diagnostic Test: Schirmer's test; Diagnostic Test: Ocular Surface Disease Index (OSDI); Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI); Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) pulse diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) constitution questionnaire; Diagnostic Test: Traditional Chinese Medicine (TCM) heart rate variability analysis; Diagnostic Test: nailfold microcirculation assessment; Diagnostic Test: iris examination; Other: Sham Laser Acupuncture
- Waiting list (Other): Group Waiting list will not receive any treatment at acupoint GB20, BL2, LI4 and LI11 twice a week 8 weeks for efficacy evaluation. And we could use the Numerical Rating Scale (NRS), Schirmer's test, Ocular Surface Disease Index (OSDI), EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI), Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, TCM constitution questionnaire, TCM heart rate variability analysis, nailfold microcirculation assessment, and iris examination for this purpose.
  Interventions: Diagnostic Test: Numerical Rating Scale (NRS); Diagnostic Test: Schirmer's test; Diagnostic Test: Ocular Surface Disease Index (OSDI); Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI); Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) pulse diagnosis; Diagnostic Test: Traditional Chinese Medicine (TCM) constitution questionnaire; Diagnostic Test: Traditional Chinese Medicine (TCM) heart rate variability analysis; Diagnostic Test: nailfold microcirculation assessment; Diagnostic Test: iris examination

INTERVENTIONS:
Other: Laser acupuncture (LA) — The RJ-Laser acupuncture device (Reimers & Janssen GmbH, Waldkirch, Germany) is used with a laser wavelength of 810 nm (infrared). The Bahr frequency B3 is set at 2398 Hz, with an energy output of 400 mW, operating in intermittent pulse mode. Each acupoint is irradiated for 15 seconds. A total of 8 bilateral acupoints are treated per session, with a total treatment time of approximately 120 seconds.
  Arms: LA+LA group of Non-SJS-DES; LA+LA group of SJS-DES; Sham+LA group of Non-SJS-DES; Sham+LA group of SJS-DES
Diagnostic Test: Numerical Rating Scale (NRS) — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the Numerical Rating Scale (NRS).
Diagnostic Test: Schirmer's test — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the Schirmer's test.
Diagnostic Test: Ocular Surface Disease Index (OSDI) — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the OSDI test.
Diagnostic Test: EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the ESSPRI.
Diagnostic Test: Traditional Chinese Medicine (TCM) tongue diagnosis — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the Traditional Chinese Medicine (TCM) tongue diagnosis.
Diagnostic Test: Traditional Chinese Medicine (TCM) pulse diagnosis — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the Traditional Chinese Medicine (TCM) pulse diagnosis.
Diagnostic Test: Traditional Chinese Medicine (TCM) constitution questionnaire — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the Traditional Chinese Medicine (TCM) constitution questionnaire.
Diagnostic Test: Traditional Chinese Medicine (TCM) heart rate variability analysis — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the Traditional Chinese Medicine (TCM) heart rate variability analysis.
Diagnostic Test: nailfold microcirculation assessment — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the nailfold microcirculation assessment.
Diagnostic Test: iris examination — LA+LA group of SJS-DES, Sham+LA group of SJS-DES, LA+LA group of Non-SJS-DES, Sham+LA group of Non-SJS-DES and Waiting list will take the iris examination.
Other: Sham Laser Acupuncture — The RJ-Laser acupuncture device (Reimers & Janssen GmbH, Waldkirch, Germany) is used with a laser wavelength of 810 nm (infrared). The Bahr frequency B3 is set at 2398 Hz, with an energy output of 400 mW, operating in intermittent pulse mode. Each acupoint is irradiated for 15 seconds. A total of 8 bilateral acupoints are treated per session, with a total treatment time of approximately 120 seconds.
  The sham laser acupuncture procedure follows the same process as the true laser acupuncture protocol, including the positioning, cleaning of acupoints, and wearing of protective goggles. However, no laser emission is delivered during the treatment. This ensures a consistent experience for the patient while maintaining the blinding integrity of the study.
  Arms: Sham+LA group of Non-SJS-DES; Sham+LA group of SJS-DES

SUMMARY:
This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the efficacy of adding laser acupuncture at Fengchi (GB20), Zanzhu (BL2), Hegu (LI4), and Quchi (LI11) acupoints to standard care for the treatment of dry eye symptoms in both Sjögren's Syndrome-related dry eye (SJS-DES) and non-Sjögren's Syndrome-related dry eye (Non-SJS-DES) populations. A total of 140 dry eye patients will be recruited and divided into two groups: 70 participants with SJS-DES and 70 with Non-SJS-DES. Participants will be randomly assigned into three groups: Sham+LA group (60 participants receiving 4 weeks of placebo laser acupuncture followed by 4 weeks of active laser acupuncture), LA+LA group (60 participants receiving 4 weeks of active laser acupuncture followed by another 4 weeks of active laser acupuncture), and a Waiting List group (20 participants receiving no laser acupuncture treatment). Each session will target the Fengchi (GB20), Zanzhu (BL2), Hegu (LI4), and Quchi (LI11) acupoints bilaterally, performed twice a week. The total study period is 8 weeks, and the treatment efficacy will be assessed at the end of the 8-week treatment. The Waiting List group (20 participants) will not receive any laser acupuncture treatment during this period. Efficacy will be evaluated using the Numerical Rating Scale (NRS), Schirmer's test, Ocular Surface Disease Index (OSDI), EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI), Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, TCM constitution questionnaire, TCM heart rate variability analysis, nailfold microcirculation assessment, and iris examination. This study aims to investigate the impact of laser acupuncture on dry eye symptom improvement and the potential markers that differentiate between SJS-DES and Non-SJS-DES patients. The goal is to develop a comprehensive integrated care model for early screening, diagnosis, and personalized treatment plans for Dry Eye Syndrome and Sjögren's Syndrome, achieving the ultimate objective of "Holistic Health Care."

DETAILED DESCRIPTION:
Method: This randomized, double-blind, placebo-controlled clinical trial aims to evaluate the efficacy of adding laser acupuncture at Fengchi (GB20), Zanzhu (BL2), Hegu (LI4), and Quchi (LI11) acupoints to standard care for the treatment of dry eye symptoms in both Sjögren's Syndrome-related dry eye (SJS-DES) and non-Sjögren's Syndrome-related dry eye (Non-SJS-DES) populations. A total of 140 dry eye patients will be recruited and divided into two groups: 70 participants with SJS-DES and 70 with Non-SJS-DES. Participants will be randomly assigned into three groups: Sham+LA group (60 participants receiving 4 weeks of placebo laser acupuncture followed by 4 weeks of active laser acupuncture), LA+LA group (60 participants receiving 4 weeks of active laser acupuncture followed by another 4 weeks of active laser acupuncture), and a Waiting List group (20 participants receiving no laser acupuncture treatment). Each session will target the Fengchi (GB20), Zanzhu (BL2), Hegu (LI4), and Quchi (LI11) acupoints bilaterally, performed twice a week. The total study period is 8 weeks, and the treatment efficacy will be assessed at the end of the 8-week treatment. The Waiting List group (20 participants) will not receive any laser acupuncture treatment during this period. Efficacy will be evaluated using the Numerical Rating Scale (NRS), Schirmer's test, Ocular Surface Disease Index (OSDI), EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI), Traditional Chinese Medicine (TCM) tongue diagnosis, TCM pulse diagnosis, TCM constitution questionnaire, TCM heart rate variability analysis, nailfold microcirculation assessment, and iris examination. This study aims to investigate the impact of laser acupuncture on dry eye symptom improvement and the potential markers that differentiate between SJS-DES and Non-SJS-DES patients. The goal is to develop a comprehensive integrated care model for early screening, diagnosis, and personalized treatment plans for Dry Eye Syndrome and Sjögren's Syndrome, achieving the ultimate objective of "Holistic Health Care."

Expected Results:

1. Assess the therapeutic differences between Sham+LA and LA+LA groups in the SJS-DES population.
2. Assess the therapeutic differences between Sham+LA and LA+LA groups in the Non-SJS-DES population.
3. Evaluate the therapeutic differences between the SJS-DES and Non-SJS-DES populations.

Keywords: Dry eye syndrome, Sjögren's syndrome, Laser Acupuncture, GB20, BL2, LI4, LI11

ELIGIBILITY:
• Dry eye syndrome

Inclusion Criteria:

1. aged between 20 and 75 years
2. Schirmer's test less than 10 mm/5 min

Exclusion Criteria:

1. Pregnancy
2. With eye inflammation or infectious eye disease
3. Accepted operation of eye

   * Sjögren's syndrome

Inclusion Criteria:

1. primary or secondary SS
2. aged between 20 and 75 years
3. fulfilled the 2002 American-European Consensus Criteria for SS (AECG)
4. had no abnormal findings of immune, liver, kidney, or blood function evaluations.

Exclusion Criteria:

1. a history of alcohol abuse, diabetes mellitus, or major life-threatening condition
2. pregnancy or breastfeeding
3. steroid pulse therapy within three months prior to the commencement of our study.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) | one year
  Numerical Rating Scale (NRS) is a tool for evaluating pain among the Dry eye syndrome (DES).
Schirmer's test | one year
  Schirmer's test is a tool for evaluating aqueous tear production among the Dry eye syndrome (DES).
Ocular Surface Disease Index (OSDI) | one year
  Ocular Surface Disease Index (OSDI) is a tool to rate the severity of dry eye disease among the Dry eye syndrome (DES).

SECONDARY OUTCOMES:
EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) | one year
  EULAR Sjögren's Syndrome Patient Reported Index (ESSPRI) is a tool for evaluating the symptoms of SJS among the Dry eye syndrome (DES).
Traditional Chinese Medicine (TCM) tongue diagnosis | one year
  Traditional Chinese Medicine (TCM) tongue diagnosis is a tool for detecting tongue expression among the Dry eye syndrome (DES).
Traditional Chinese Medicine (TCM) pulse diagnosis | one year
  Traditional Chinese Medicine (TCM) pulse diagnosis is a tool for detecting tongue expression pulse pattern among the Dry eye syndrome (DES).
Traditional Chinese Medicine (TCM) constitution questionnaire | one year
  Traditional Chinese Medicine (TCM) constitution questionnaire is a tool for detecting the constitution among the Dry eye syndrome (DES).
Traditional Chinese Medicine (TCM) heart rate variability analysis | one year
  Traditional Chinese Medicine (TCM) heart rate variability analysis is a tool for detecting ratio between High-frequency (HF) activity and low-frequency (LF) activity among the Dry eye syndrome (DES).
Nailfold microcirculation assessment | one year
  Nailfold microcirculation assessment is a tool for detecting the status of nailfold microcirculation among the Dry eye syndrome (DES).
Iris examination | one year
  Iris examination is a tool for detecting the status of iris among the Dry eye syndrome (DES).

CONTACTS AND LOCATIONS:
Locations (1):
- Ching-Mao Chang, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
The decision to share individual participant data (IPD) is currently undecided due to ongoing discussions regarding data management, privacy concerns, and compliance with institutional and regulatory requirements. Additional considerations include the establishment of appropriate data-sharing agreements, ensuring participant confidentiality, and defining the scope and method of data access. Once these factors are thoroughly evaluated and addressed, a final decision regarding IPD sharing will be made in accordance with ethical guidelines and applicable regulations.